CLINICAL TRIAL: NCT06837467
Title: Differential Expression of SERCA and Myosin Heavy Chain Isoforms in Rat Laryngeal Muscles
Brief Title: Differential SERCA Expression in Laryngeal Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Elrabie Ahmed, Clinical Professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: sohag-5-24-2023-01
Record Dates: First submitted 2025-02-07; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Myopathy
Keywords: SERCA and MHC isoform
MeSH Terms: conditions — Muscular Diseases | interventions — Immunohistochemistry

STUDY DESIGN:
Intervention Model Description: In this study, male adult Wistar rats (Shimizu Laboratory Supplies Co., Kyoto, Japan), 8-12 weeks of age, weighing 280-350 g (N=10) were used as young rats. In addition, 24-month-old rats (N=10) were employed as aged models.
  In 8-12 weeks, aged rats, the larynx was approached through a midline incision using a standard operating microscope under anesthesia with sodium pentobarbital. After identification of the right recurrent and superior laryngeal nerves, a 1 cm segment was removed from the right recurrent laryngeal nerve and both ends were ligated. The right superior laryngeal nerve was also divided. The denervated rat groups were sacriﬁced after 2, 4, 8, and 12 weeks. The larynx was collected and prepared for IHC using the same procedure described above (n = 5 in each group).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young rat (Experimental): male adult Wistar rats (Shimizu Laboratory Supplies Co., Kyoto, Japan), 8-12 weeks of age, weighing 280-350 g (N=10) were used as young rats Immunohistochemistry (IHC) with anti-SERCA1 or -SERCA2 and anti-MHC I or -MHCII (Table 1) antibodies for 1-2 days at 4 ◦C, then washed and incubated with Alexa Fluor® 488 donkey anti-mouse IgG and Fluor® 594 donkey anti-goat IgG secondary Abs for 1 hour at room temperature. Double IHC was performed using (anti-SERCA1 + anti-SERCA2) and (anti-SERCA2 + anti-MHCII) combinations to check co-expression. In double IHC, the same steps were done as before with mixture of primary or secondary antibodies with same dilutions.
  Interventions: Diagnostic Test: Immunohistochemistry (IHC)
- old rats (Experimental): 24-month-old rats (N=10) were employed as aged models. Immunohistochemistry (IHC) with anti-SERCA1 or -SERCA2 and anti-MHC I or -MHCII (Table 1) antibodies for 1-2 days at 4 ◦C, then washed, and incubated with Alexa Fluor® 488 donkey anti-mouse IgG and Fluor® 594 donkey anti-goat IgG secondary Abs for 1 hour at room temperature. Double IHC was performed using (anti-SERCA1 + anti-SERCA2) and (anti-SERCA2 + anti-MHCII) combinations to check co-expression. In double IHC, the same steps were done as before with mixture of primary or secondary antibodies with same dilutions.
  Interventions: Diagnostic Test: Immunohistochemistry (IHC)
- Denervated rats (Active Comparator): In 8-12 weeks, aged rats, the larynx was approached through a midline incision using a standard operating microscope under anesthesia with sodium pentobarbital. After identification of the right recurrent and superior laryngeal nerves, a 1 cm segment was removed from the right recurrent laryngeal nerve and both ends were ligated. The right superior laryngeal nerve was also divided. The denervated rat groups were sacriﬁced after 2, 4, 8, and 12 weeks. The larynx was collected and prepared for IHC using the same procedure described above (n = 5 in each group).
  Immunohistochemistry (IHC) with anti-SERCA1 or -SERCA2 and anti-MHC I or -MHCII (Table 1) antibodies for 1-2 days at 4 ◦C, then washed, and incubated with Alexa Fluor® 488 donkey anti-mouse IgG and Fluor® 594 donkey anti-goat IgG secondary Abs for 1 hour at room temperature. Double IHC was performed using (anti-SERCA1 + anti-SERCA2) and (anti-SERCA2 + anti-MHCII) combinations to check co-expression. In double IHC.
  Interventions: Diagnostic Test: Immunohistochemistry (IHC)

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry (IHC) — We faced unsuccessful fast fiber type's identification on frozen sections then we shifted to paraffin sections. Deparaffinized sections were incubated with 3% H2O2 in PBS for 10 minutes followed by microwave treatment (5 minutes ×3 times at 500 Watt in citrate buffer, pH 6). Then, sections were incubated in blocking solution (0.3 M glycine, 50 mM ammonium chloride, and 1% BSA in PBS) for 30 minutes before incubation in primary antibodies. Sections were incubated with anti-SERCA1 or -SERCA2 and anti-MHC I or -MHCII (Table 1) antibodies for 1-2 days at 4 ◦C, then washed, and incubated with Alexa Fluor® 488 donkey anti-mouse IgG and Fluor® 594 donkey anti-goat IgG secondary Abs for 1 hour at room temperature. Double IHC was performed using (anti-SERCA1 + anti-SERCA2) and (anti-SERCA2 + anti-MHCII) combinations to check co-expression. In double IHC, the same steps were done as before with mixture of primary or secondary antibodies with same dilutions.

SUMMARY:
Immuno-localization of SERCA and MHC isoform (SERCA1, SERCA2, MHC I, and MHCII) expression and co-expression in the five ILMs were investigated in both young and aged rats with immunohistochemistry. Special concern has been placed to the denervation effect on ILMS.

DETAILED DESCRIPTION:
Animals In this study, male adult Wistar rats (Shimizu Laboratory Supplies Co., Kyoto, Japan), 8-12 weeks of age, weighing 280-350 g (N=10) were used as young rats. In addition, 24-month-old rats (N=10) were employed as aged models.

Animal tissue preparation Animals were anesthetized with an intraperitoneal injection of sodium pentobarbital (dose 30-60 mg/kg) and were fixed with 4% paraformaldehyde following cardiac perfusion with 0.01 M phosphate-buffered saline (PBS). The larynges were excised immediately and immersed in the same fixative for approximately 12 hours at (4°C). Tissues were processed in paraffin and sectioned using a microtome (8-10 μm thickness).

The intrinsic laryngeal muscles studied were: 1) medial and lateral thyroarytenoid (MTA, LTA), (2) lateral cricoarytenoid (LCA), (3) Superior cricoarytenoid (SCA), (4) posterior cricoarytenoid (PCA), and (5) cricothyroid (CT).

Immunohistochemistry (IHC) The investigators faced unsuccessful fast fiber type identification on frozen sections then we shifted to paraffin sections. Deparaffinized sections were incubated with 3% H2O2 in PBS for 10 minutes followed by microwave treatment (5 minutes ×3 times at 500 Watt in citrate buffer, pH 6). Then, sections were incubated in a blocking solution (0.3 M glycine, 50 mM ammonium chloride, and 1% BSA in PBS) for 30 minutes before incubation in primary antibodies. Sections were incubated with anti-SERCA1 or -SERCA2 and anti-MHC I or -MHCII (Table 1) antibodies for 1-2 days at 4 ◦C, then washed, and incubated with Alexa Fluor® 488 donkey anti-mouse IgG and Fluor® 594 donkey anti-goat IgG secondary Abs for 1 hour at room temperature. Double IHC was performed using (anti-SERCA1 + anti-SERCA2) and (anti-SERCA2 + anti-MHCII) combinations to check co-expression. In double IHC, the same steps were done with a mixture of primary or secondary antibodies with the same dilutions.

Immunostained tissue sections were examined using a FV-1000 laser confocal microscope (Olympus, Tokyo, Japan). ImageJ 1.46 software was used to manually count and calculate the percentage of positive cells for each antibody.

Immunohistochemistry for denervated rat In 8-12 weeks, aged rats, the larynx was approached through a midline incision using a standard operating microscope under anesthesia with sodium pentobarbital. After identification of the right recurrent and superior laryngeal nerves, a 1 cm segment was removed from the right recurrent laryngeal nerve and both ends were ligated. The right superior laryngeal nerve was also divided. The denervated rat groups were sacriﬁced after 2, 4, 8, and 12 weeks. The larynx was collected and prepared for IHC using the same procedure described above (n = 5 in each group).

MHC subtypes using multi-color fiber typing:

At the beginning of our research, we tried the frozen section. After trials of several techniques to decrease autofluorescence and background noise, the investigators failed to have good staining. Then, the investigators discontinued MHC subtyping and shifted to paraffin-embedded blocks Statistical analysis The relative SERCA and MHC composition for each muscle was calculated. The available data for the positive cell percentage of each rat antibody were statistically analyzed using SPSS statistical software, version 16. Statistical comparisons were performed using the unpaired two-tailed Student's t-test and were considered significant at P < 0.05.

One-way analysis of variance (ANOVA) followed by Scheffe's post hoc test was performed to compare the MHC and SERCA composition for each muscle in denervation with the contralateral side and young with age. Values presented are means ± SD (standard deviation), with SD being across rats.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 weeks of age, weighing 280-350 g (N=10) were used as young rats. In addition, 24-month-old rats (N=10) were employed as aged models.

Exclusion Criteria:

-

Ages: 8 Weeks to 24 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Immuno-localization of SERCA and MHC isoform | 6 months
  Immuno-localization of SERCA and MHC isoform (SERCA1, SERCA2, MHC I, and MHCII) expression and co-expression in the five ILMs

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Ahmed, Study Director — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao VH, Abaza M, Spiegel JR, Mandel S, Hawkshaw M, Heuer RJ, Sataloff RT. Laryngeal myasthenia gravis: report of 40 cases. J Voice. 2001 Mar;15(1):122-30. doi: 10.1016/S0892-1997(01)00012-1. PMID 12269627
- [Background] Marques MJ, Ferretti R, Vomero VU, Minatel E, Neto HS. Intrinsic laryngeal muscles are spared from myonecrosis in the mdx mouse model of Duchenne muscular dystrophy. Muscle Nerve. 2007 Mar;35(3):349-53. doi: 10.1002/mus.20697. PMID 17143878